CLINICAL TRIAL: NCT02033590
Title: Clinical and Economic Outcomes With the Use of SERI® Surgical Scaffold in Direct-to-implant Breast Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Strategic priorities impacted study
Sponsor: Sofregen Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURE-005
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Breast Reconstruction

ARMS (1):
- SERI® Surgical Scaffold (Experimental)
  Interventions: Device: Biodegradable (purified) surgical silk scaffold

INTERVENTIONS:
Device: Biodegradable (purified) surgical silk scaffold

SUMMARY:
The objective of this study is to prospectively observe clinical and economic outcomes with the use of SERI® in direct-to-implant breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to undergo immediate breast reconstruction following a skin-sparing or nipple sparing mastectomy with healthy, sufficiently thick, well-vascularized skin flaps, and the implantation of SERI® Surgical Scaffold and breast implant
* Be female, between 18 and 65 years of age at the time of enrollment

Exclusion Criteria:

* Have undergone prior radiation treatment on the study breast(s) and/or is preoperatively evaluated to require radiation treatment to the study breast(s) during the course of the study
* Have undergone a skin reducing mastectomy
* Have a BMI that is <17 or ≥ 30
* Predicted implant weight more than 500 grams
* Have a known allergy to silk
* Have an abscess or active infection at any location within one month prior to surgery
* Be pregnant, lactating, or if of childbearing potential, be unwilling to use contraceptive methods and avoid pregnancy throughout the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate of implant loss (SERI® and breast implant) | 52 weeks